CLINICAL TRIAL: NCT02528643
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Enzalutamide in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: A Study to Assess the Efficacy and Safety of Enzalutamide in Subjects With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9785-CL-3021; 2014-004283-37 (EudraCT Number)
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: MDV3100; advanced hepatocellular carcinoma; enzalutamide; Xtandi; ASP9785
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enzalutamide 160 mg (Experimental): Participants received enzalutamide 160 milligrams (mg) capsules, orally QD during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Eligible participants received enzalutamide 160 mg capsules, orally QD during open label period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
  Interventions: Drug: Enzalutamide
- Placebo (Placebo Comparator): Participants received enzalutamide matching placebo orally, once daily (QD) during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enzalutamide — Oral capsule
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide 160 mg
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy of enzalutamide in participants with advanced hepatocellular carcinoma (HCC) as measured by overall survival (OS).

This study also evaluated the safety of enzalutamide; pharmacokinetics of enzalutamide and the active metabolite N-desmethyl and Progression Free Survival (PFS) of enzalutamide as compared to placebo in participants with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age or is considered an adult according to local regulation at the time of signing informed consent.
* Subject has a documented diagnosis of advanced HCC of any etiology.
* Subject has BCLC stage B or C.
* Subject's lesions are not amenable to local therapies which may be beneficial, such as transarterial chemoembolization (TACE), radiofrequency ablation, radiotherapy, etc., and the subject is not a candidate for any curative treatments such as resection or liver transplant.
* Subject has hepatic function status of Child Pugh Class A at Screening.
* Subject received prior systemic treatment for HCC with sorafenib or other anti-VEGF therapy and had confirmed disease progression or discontinued treatment due to a drug-related toxicity. Subject may have received 1 line of systemic therapy before or after sorafenib/anti-VEGF treatment.
* Subject has adequately recovered from toxicities due to prior HCC therapy to ≤ grade 1.
* Subject has an ECOG performance status ≤ 1 at Screening and on Day 1.
* Subject has available formalin-fixed, paraffin-embedded tumor specimen with adequate viable tumor cells in a tissue block or unstained serial slides accompanied by an associated pathology report prior to enrollment. Archival or fresh biopsy tissue is required.
* Subject has an estimated life expectancy of at least 3 months on Day 1, in the opinion of the investigator.
* Female subject is either:

  * Not of childbearing potential: postmenopausal (defined as no spontaneous menses for at least 12 consecutive months prior to Screening with follicle-stimulating hormone [FSH] > 40 IU/L for women < 55 years of age at Screening), or documented to be surgically sterile or status posthysterectomy (at least 1 month prior to Screening).
  * Or, if of childbearing potential: must have a negative urine pregnancy test at Screening and on Day 1 before the first dose of study drug is administered, and must use 2 acceptable methods of birth control* if sexually active from Screening through 3 months after the last dose of study drug.
* Sexually active male subject and his female partner who is of childbearing potential must use 2 acceptable methods of birth control from Screening through 3 months after the last dose of study drug.

  * Two acceptable methods of birth control are as follows:
  * Condom (barrier method of contraception); AND
  * One of the following is required: Placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female subject or female partner of a male subject; Additional barrier method: contraceptive sponge or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female subject or female partner of a male subject. For male subject or male partner of female subject, vasectomy or other procedure resulting in infertility (e.g., bilateral orchiectomy) performed at least 6 months before Screening. Tubal ligation in the female partner of a male subject performed at least 6 months before Screening. Established and ongoing use of oral, injected, or implanted hormonal contraceptive by female partner of a male subject.
* Female subject must not be breastfeeding at Screening or during the study period and for 3 months after final study drug administration.
* Subject must agree not to donate sperm or ova from first dose of study drug through 3 months after the last dose of study drug.
* Throughout the study, male subject must use a condom if having sex with a pregnant woman.
* Subject must be able to swallow study drug and comply with study requirements.
* Subject agrees not to participate in another interventional study while on treatment.
* Received double-blind enzalutamide study treatment during the main study.

Exclusion Criteria:

* Subject has a severe concurrent disease, infection or comorbidity that, in the judgment of the investigator, would make the subject inappropriate for enrollment.
* Subject has fibrolamellar variant of HCC.
* Subject has status of Child-Pugh Class B or C at Screening.
* Subject has a history of organ allograft including liver transplant.
* Subject has uncontrolled symptomatic ascites.
* Subject has known or suspected brain metastasis or active leptomeningeal disease.
* Subject has a history of a non-HCC malignancy with the following exceptions:

  * The subject with a previous history of a noninvasive carcinoma is eligible if in the opinion of the investigator he/she has had successful curative treatment any time prior to Screening and requires no further therapy for the malignancy.
  * For all other malignancies, the subject is eligible if he/she has undergone potentially curative therapy and has been considered disease free for at least 3 years prior to Screening.
* Subject has inadequate marrow, hepatic, and/or renal function at the Screening Visit defined as:

  * Absolute neutrophil count < 1.5 x109/L (< 1500 cells/mm3)
  * Platelet count < 50 x109/L (< 50,000 cells/mm3)
  * Hemoglobin < 8.5 g/dL (< 5.3 mmol/L)
  * International normalized ratio > 1.7
  * Albumin < 2.8 g/dL (< 28 g/L)
  * Total bilirubin (TBL) > 2 x ULN
  * AST or ALT > 5 x ULN
  * Creatinine > 1.5 x ULN
  * Note: Transfusions/infusions to meet eligibility criteria are not allowed but if in the opinion of the Principal Investigator, it is beneficial, the patient may be rescreened after receiving one of these procedures.
* Subject has a history of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma, encephalopathy within 3 months of Day 1).
* Subject has a history of bleeding esophageal varices within 3 months before the Day 1 visit.
* Subject has a history of loss of consciousness or transient ischemic attack within 12 months before the Day 1 visit.
* Subject has clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months before the Day 1 visit.
  * Uncontrolled angina within 6 months before the Day 1 visit.
  * Congestive heart failure New York Heart Association (NYHA) Class III or IV or history of congestive heart failure NYHA Class III or IV in the past, unless a Screening echocardiogram or multi-gated acquisition scan performed within 3 months before the Day 1 visit reveals a left ventricular ejection fraction that is ≥ 45%.
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, Torsade de Pointes).
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place.
  * Hypotension as indicated by systolic blood pressure < 86 mmHg on 2 consecutive measurements at the Screening visit.
  * Bradycardia (in the presence of known cardiovascular disease) as indicated by a heart rate of < 50 beats per minute on the Screening electrocardiogram (ECG) recording.
  * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg on 2 consecutive measurements at the Screening visit.
* Subject has a gastrointestinal disorder affecting absorption.
* Subject had previous local therapy (e.g., surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation) within 14 days prior to Day 1, has not recovered from toxicities from prior local therapy or may require major surgical procedure during the course of the study.
* Subject has received chemotherapy, immunotherapy or any other systemic anticancer therapy (including sorafenib) or any other investigational drug within 14 days prior to the Day 1 visit.
* Subject has received an agent that either blocks androgen synthesis or targets the AR (e.g., abiraterone acetate, bicalutamide, enzalutamide, ARN-509 or other investigational AR signaling inhibitors). The exception of spironolactone is allowed after Medical Monitor consultation.
* Subject has used any of the following within 28 days before the Day 1 visit:

  * 5-α reductase inhibitors
  * Systemic androgens and estrogens (vaginal estrogen creams are allowed)
  * Herbal therapies, with an antitumor effect.
* Subject has a known history of positive test for Human Immunodeficiency Virus.
* Subject has shown a hypersensitivity reaction to the active pharmaceutical ingredient or any of the enzalutamide capsule components, including caprylocaproyl polyoxylglycerides (Labrasol), butylated hydroxyanisole and butylated hydroxytoluene.
* Subject has addictive/substance abuse problems.
* Subject has any other condition or reason that, in the opinion of the investigator, interferes with the ability of the subject to participate in the trial, places the subject at undue risk or complicates the interpretation of safety data.
* Received double-blind placebo during the main study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (38):
- United States (8):
  - Site US10003, San Francisco, California
  - Site US10009, Skokie, Illinois
  - Site US10017, Minneapolis, Minnesota
  - Site US10021, Lebanon, New Hampshire
  - Site US10008, Portland, Oregon
  - Site US10014, Philadelphia, Pennsylvania
  - Site US10019, Philadelphia, Pennsylvania
  - Site US10016, Milwaukee, Wisconsin
- Canada (3):
  - Site CA15001, Toronto, Ontario
  - Site CA15002, Montreal, Quebec
  - Site CA15003, Montreal
- Hong Kong (2):
  - Site HK85202, Kowloon
  - Site HK85204, Shatin
- Italy (6):
  - Site IT39008, Rozzano, Milan
  - Site IT39005, Benevento
  - Site IT39002, Milan
  - Site IT39006, Milan
  - Site IT39011, Padua
  - Site IT39004, Pavia
- Site US10001, San Juan, Puerto Rico
- South Korea (6):
  - Site KR82002, Seongnam-si, Gyeonggi-do
  - Site KR82005, Seoul, Seoul Teugbyeolsi
  - Site KR82006, Seoul
  - Site KR82007, Seoul
  - Site KR82004, Seoul
  - Site KR82001, Seoul
- Spain (3):
  - Site ES34003, Barcelona
  - Site ES34006, Córdoba
  - Site ES34004, Madrid
- Taiwan (4):
  - Site TW88603, Douliu
  - Site TW88606, Tainan
  - Site TW88605, Tainan
  - Site TW88604, Taipei
- United Kingdom (5):
  - Site GB44007, Birmingham
  - Site GB44004, London
  - Site GB44008, London
  - Site GB44005, Manchester
  - Site GB44002, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Ryoo BY, Palmer DH, Park SR, Rimassa L, Debashis Sarker, Daniele B, Steinberg J, Lopez B, Lim HY. Efficacy and Safety Results from a Phase 2, Randomized, Double-Blind Study of Enzalutamide Versus Placebo in Advanced Hepatocellular Carcinoma. Clin Drug Investig. 2021 Sep;41(9):795-808. doi: 10.1007/s40261-021-01063-0. Epub 2021 Aug 5. PMID 34351608
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/?pid=9785-CL-3021
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14696&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 37 sites in 9 countries in Europe, Asia, and North America. Participants with hepatocellular carcinoma (HCC) of any etiology whose disease had progressed on or who were intolerant to sorafenib or other antivascular endothelial growth factor (VEGF) therapy in the advanced setting were enrolled.
  Double blind treatment (DB) Open label (OL).
Pre-assignment Details: Eligible participants were stratified by geographic region (Asia vs other) and Eastern Cooperative Oncology Group (ECOG) performance (0 vs 1) and randomized in a 2:1 ratio. Participants who discontinued treatment entered a follow-up period
  .
Groups:
- Enzalutamide: Participants received enzalutamide 160 milligrams (mg) capsules, orally QD during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Eligible participants received enzalutamide 160 mg capsules, orally QD during open label period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
Period: DB (Median Duration up to 14.65 Months)
Arm/Group | Placebo | Enzalutamide
Started | 55 | 110
Treated | 55 | 107
Completed | 0 | 0
Not Completed | 55 | 110
Not completed — Adverse Event | 5 | 8
Not completed — Death | 1 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Progressive Disease | 44 | 82
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Miscellaneous | 3 | 5
Period: OL (Median Duration up to 27.56 Months)
Arm/Group | Placebo | Enzalutamide
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomized participants regardless of whether or not participants received study drug.
Groups:
- Placebo: Participants received enzalutamide matching placebo orally, QD during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
- Enzalutamide: Participants received enzalutamide 160 mg capsules, orally QD during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Enzalutamide | Total
Number analyzed (Participants) | 55 | 110 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (12.5) | 63.7 (10.9) | 63.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 21
  Male | 49 | 95 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 55 | 107 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 52 | 78
  Black or African American | 3 | 5 | 8
  Asian | 25 | 52 | 77
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 1 | 0 | 1
Geographic Region [Count of Participants; unit: Participants]
  Asia | 24 | 48 | 72
  Other | 31 | 62 | 93
Eastern Cooperative Oncology Group (ECOG) PS (0,1) [Number; unit: Participants] — ECOG PS was measured on 6 point scale 0-Fully active, able to carry on all pre-disease performance without restriction 1- Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature 2-Ambulatory & capable of all self-care but unable to carry out any work activities Up & about more than 50% of waking hours 3-Capable of only limited self-care, confined to bed or chair more than 50% of waking hours 4-Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair 5-Dead Participants were categorized based on ECOGPS 0 or 1
  Participants
    ECOG PS = 0 | 23 | 43 | 66
    ECOG PS = 1 | 32 | 67 | 99

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the documented date of death from any cause. Participants who were still alive at the time of the data cut-off date was censored on the last date known to be alive or at the data cutoff date, whichever occurs first. Results based on Kaplan-Meier estimates.
Time Frame: From date of randomization up to data cut-off date 02 Oct 2017 (approximately 22 months); median follow-up time was 14.65 months for enzalutamide and 13.83 for placebo.
Population: The analysis population was the FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Enzalutamide
Number analyzed (Participants) | 55 | 110
months | 7.69 [5.82 to 13.77] | 7.75 [6.05 to 9.92]
Statistical Analysis 1: Comparison: Placebo vs Enzalutamide; Stratified Analysis. The null hypothesis was stated as: OS distributions of the 2 arms are equivalent. The alternative hypothesis was stated as: OS is prolonged in enzalutamide arm. The null hypothesis was tested using a stratified one-sided log-rank test at the 0.10 level. Stratification factors were ECOG performance status and region from eCRF; Test type: Superiority; p = 0.248, Log Rank — One-sided p-value; Hazard Ratio (HR) = 1.146, 95% CI 2-sided [0.774 to 1.696] — Calculated using a Cox proportional hazard model, stratified by geographic region and ECOG performance status. Hazard ratio < 1 indicated a reduction in hazard rate in favor of enzalutamide group
Statistical Analysis 2: Comparison: Placebo vs Enzalutamide; Unstratified Analysis. The null hypothesis was stated as: OS distributions of the 2 arms are equivalent. The alternative hypothesis was stated as: OS is prolonged in enzalutamide arm. The null hypothesis was tested using a one-sided log-rank test at the 0.10 level; Test type: Superiority; p = 0.252, Log Rank — One-sided p-value; Hazard Ratio (HR) = 1.142, 95% CI 2-sided [0.773 to 1.688] — Calculated using a Cox proportional hazard model. Hazard ratio < 1 indicated a reduction in hazard rate in favor of enzalutamide group

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety was assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A treatment-emergent AE (TEAE) was defined as an AE observed after starting administration of the study drug up to 30 days after last dose of study drug or initiation of new treatment, whichever comes first. AEs were considered as serious if resulted in in death, was life-threatening resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly or birth defect, required inpatient hospitalization or led to prolongation of hospitalization and other medically important events.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug median (minimum, maximum) treatment duration was 64.0 (6, 1736) days for enzalutamide and 64.0 (12, 490) for placebo
Population: The analysis population was the safety analysis set (SAF), which consisted of all participants who have received at least 1 or partial capsule of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Enzalutamide: Participants received enzalutamide 160 milligrams (mg) capsules, orally, QD during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Eligible participants received enzalutamide 160 mg capsules, orally QD during open label period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
Arm/Group | Placebo | Enzalutamide
Number analyzed (Participants) | 55 | 107
Participants
  TEAE | 50 | 105
  Drug-related TEAEs | 24 | 69
  Deaths | 45 | 82
  TEAE Leading to Death | 6 | 12
  Drug-related TEAEs Leading to Death | 0 | 0
  Serious TEAEs | 22 | 47
  Drug-related Serious TEAEs | 3 | 7
  TEAEs Leading to Treatment Withdrawal | 14 | 34
  Drug-related TEAEs Leading to Treatment Withdrawal | 4 | 7

3. Secondary Outcome: Plasma Trough Concentrations of Enzalutamide
Description: Blood samples were collected for analysis.
Time Frame: Predose at weeks 5, 9 and 13
Population: The analysis population was the pharmacokinetics analysis set (PKAS), consisted of the subset of the SAF population for whom at least 1 quantifiable enzalutamide and N-desmethyl enzalutamide concentration value was available. Participants who had available concentration data were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 96
μg/mL
  Week 5: number analyzed (Participants) | 66
  Week 5 | 14.29 (4.15)
  Week 9: number analyzed (Participants) | 40
  Week 9 | 12.15 (4.68)
  Week 13: number analyzed (Participants) | 36
  Week 13 | 12.45 (5.44)

4. Secondary Outcome: Plasma Trough Concentrations N-desmethyl Enzalutamide (M2 Metabolite)
Description: Blood samples were collected for analysis.
Time Frame: Predose at weeks 5, 9 and 13
Population: The analysis population was the PKAS, with participants who had available concentration data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 96
μg/mL
  Week 5: number analyzed (Participants) | 66
  Week 5 | 11.01 (3.63)
  Week 9: number analyzed (Participants) | 40
  Week 9 | 12.65 (3.89)
  Week 13: number analyzed (Participants) | 36
  Week 13 | 12.21 (4.94)

5. Secondary Outcome: Plasma Trough Concentrations of MDPC0001 (M1 Metabolite)
Description: Blood samples were collected for analysis.
Time Frame: Predose at weeks 5, 9 and 13
Population: The analysis population was the PKAS, with participants who had available concentration data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 96
μg/mL
  Week 5: number analyzed (Participants) | 66
  Week 5 | 4.70 (3.86)
  Week 9: number analyzed (Participants) | 40
  Week 9 | 5.60 (5.63)
  Week 13: number analyzed (Participants) | 36
  Week 13 | 6.12 (4.24)

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the date of documented radiographic disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the investigator or death from any cause on study, whichever occurred first. The earliest of the censoring times was used: Participants with (1) no evaluable postbaseline imaging assessments or did not die were censored at the randomization date; (2) no radiographical progression or did not die before analysis cutoff date were censored at the last radiological assessment date before analysis cutoff date; (3) with no radiographical progression or did not die before new HCC treatment was censored at the last radiological assessment date before start of new HCC treatment. Based on Kaplan-Meier.
Time Frame: as for outcome 1
Population: The analysis population was the FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Enzalutamide
Number analyzed (Participants) | 55 | 110
months | 1.87 [1.84 to 3.45] | 2.23 [1.87 to 3.52]
Statistical Analysis 1: Comparison: Placebo vs Enzalutamide; Stratified Analysis. The null hypothesis was stated as: PFS distributions of the 2 arms are equivalent. The alternative hypothesis was stated as: PFS is prolonged in enzalutamide arm. The null hypothesis was tested using a stratified one-sided log-rank test at the 0.10 level. Stratification factors were ECOG performance status and region from eCRF; Test type: Superiority; p = 0.396, Log Rank — One-sided p-value; Hazard Ratio (HR) = 1.039, 95% CI 2-sided [0.732 to 1.474] — Calculated using a Cox proportional hazard model, stratified by ECOG performance status and region. Hazard ratio < 1 indicated a reduction in hazard rate in favor of enzalutamide group
Statistical Analysis 2: Comparison: Placebo vs Enzalutamide; Unstratified Analysis. The null hypothesis was stated as: PFS distributions of the 2 arms are equivalent. The alternative hypothesis was stated as: PFS is prolonged in enzalutamide arm. The null hypothesis was tested using a one-sided log-rank test at the 0.10 level; Test type: Superiority; p = 0.586, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.959, 95% CI 2-sided [0.684 to 1.345] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30days after last dose of study drug median (minimum, maximum) treatment duration was 64.0 (6, 1736) days for enzalutamide and 64.0 (12, 490) for placebo
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg capsules, orally, QD during double blind treatment period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Eligible participants received enzalutamide 160 mg capsules, orally QD during open label period until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. Median treatment duration was 64 days.
Arm/Group | Placebo | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 45/55 | 82/107
Serious Adverse Events (participants affected / at risk) | 22/55 | 47/107
Other Adverse Events (participants affected / at risk) | 46/55 | 96/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | Enzalutamide (N=107)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (8)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 5 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (4)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (4)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 14 (20)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | Enzalutamide (N=107)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 12 (17)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (6) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 15 (24)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 7 (10)
Ascites (Gastrointestinal disorders) | 2 (2) | 11 (16)
Constipation (Gastrointestinal disorders) | 5 (5) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 13 (22) | 13 (17)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 9 (13)
Nausea (Gastrointestinal disorders) | 6 (6) | 29 (33)
Vomiting (Gastrointestinal disorders) | 5 (5) | 11 (13)
Asthenia (General disorders) | 11 (12) | 11 (26)
Fatigue (General disorders) | 10 (11) | 38 (49)
Oedema peripheral (General disorders) | 3 (3) | 6 (7)
Pyrexia (General disorders) | 5 (5) | 8 (9)
Alanine aminotransferase increased (Investigations) | 7 (10) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 9 (10) | 16 (23)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 5 (5)
Blood bilirubin increased (Investigations) | 2 (2) | 6 (9)
Weight decreased (Investigations) | 5 (6) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 33 (40)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (8) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Dizziness (Nervous system disorders) | 5 (7) | 4 (7)
Dysgeusia (Nervous system disorders) | 4 (5) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 7 (9)
Insomnia (Psychiatric disorders) | 7 (7) | 13 (14)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 12 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 13 (14)
Hypertension (Vascular disorders) | 0 (0) | 6 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT02528643/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT02528643/SAP_001.pdf